CLINICAL TRIAL: NCT03586934
Title: Multimodal Anesthesia and Analgesia for Total Shoulder and Reverse Total Shoulder Arthroplasty: A Randomized Controlled Trial
Brief Title: Multimodal Analgesia in Shoulder Arthroplasty
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficult to enroll patients for the study
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORA 17071004
Record Dates: First submitted 2018-06-27; First posted 2018-07-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Shoulder Pain; Opioid Use
MeSH Terms: conditions — Shoulder Pain | interventions — Acetaminophen; Celecoxib; Ropivacaine; Ketorolac; Ketorolac Tromethamine; Oxycodone; Tramadol; Morphine; Hydrocodone; oxycodone-acetaminophen; Meloxicam

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional (Standard) Protocol (Other): Preoperative Single shot interscalene block (30 mL 0.5 ropivacaine), postoperative morphine patient controlled analgesia (1 mg/10 min/30 mg) with Hydrocodone-Acetaminophen (oral, 5/325 mg, 1 tab q4h pro re nata (PRN) for pain score of 1-3), Hydrocodone-Acetaminophen (oral, 10/325 mg, 1 tab q4h PRN for pain score of 4-6) Morphine injectable solution (2 mg IV q3h PRN for pain score 7-10), and oxycodone hydrochloride (oral, 10 mg q12h x2 doses) through postoperative day one. Discharged from hospital with hydrocodone bitartrate and acetaminophen (Norco) (5/325 mg or 10/325 mg, 1-2 oral tabs q4-6h PRN pain) script.
  Interventions: Drug: Ropivacaine; Drug: Morphine Injectable Solution; Drug: hydrocodone bitartrate and acetaminophen; Drug: Morphine; Drug: Oxycodone Hydrochloride
- Multimodal Anesthesia and Analgesia (Experimental): Under age 75: Preop: acetaminophen 1000 mg oral, celecoxib 400 mg oral. Interscalene block (30 ml 0.5% ropivacaine with 1:200,000 epinephrine). Intraop: ketorolac 15 mg IV, acetaminophen injectable product. Postop: acetaminophen 500 mg oral, oxycontin 10 mg oral. Breakthrough: ketorolac 15 mg IV, oxycodone 10 mg oral. Floor: tramadol 100 mg q6h oral, acetaminophen 1 g q8h oral, celecoxib 200 mg q12h oral, ketorolac 15 mg IV q6h. Breakthrough: Pain scores 4-6: oxycodone 5 mg q4h PRN oral, pain scores 7-10: oxycodone 10 mg q4h PRN oral. Discharge: acetaminophen 1 g q8h oral, tramadol 100 mg q8h oral, celecoxib 200 mg q12h oral or meloxicam 15 mg daily oral, oxycodone 5 mg q4h PRN oral.
  75 or older: Same except: Preop: celecoxib 200 mg oral. PACU meds: acetaminophen 500 mg oral. No OxyER.
  Interventions: Drug: Acetaminophen; Drug: Celecoxib 200mg; Drug: Celecoxib 400 mg; Drug: Ropivacaine; Drug: Ketorolac; Drug: Acetaminophen Injectable Product; Drug: Oxycodone; Drug: Tramadol; Drug: Meloxicam

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen Tablet
  Other Names: Tylenol
  Arms: Multimodal Anesthesia and Analgesia
Drug: Celecoxib 200mg — Celecoxib Tablet
  Other Names: Celebrex
  Arms: Multimodal Anesthesia and Analgesia
Drug: Celecoxib 400 mg — Celecoxib Tablet
  Other Names: Celebrex
  Arms: Multimodal Anesthesia and Analgesia
Drug: Ropivacaine — Ropivicaine nerve block (injection)
Drug: Ketorolac — ketorolac injection
  Other Names: Toradol
  Arms: Multimodal Anesthesia and Analgesia
Drug: Acetaminophen Injectable Product — Acetaminophen injection
  Other Names: Tylenol
  Arms: Multimodal Anesthesia and Analgesia
Drug: Oxycodone — oxycodone tablet
  Other Names: OxyIR
  Arms: Multimodal Anesthesia and Analgesia
Drug: Tramadol — Tramadol tablet
  Other Names: Ultram
  Arms: Multimodal Anesthesia and Analgesia
Drug: Morphine Injectable Solution — Morphine Patient Controlled Analgesia
  Other Names: Morphine
  Arms: Traditional (Standard) Protocol
Drug: hydrocodone bitartrate and acetaminophen — Norco tablet
  Other Names: Norco
  Arms: Traditional (Standard) Protocol
Drug: Morphine — morphine injection
  Arms: Traditional (Standard) Protocol
Drug: Oxycodone Hydrochloride — oxycodone hydrochloride tablet
  Other Names: Oxycontin; OxyER
  Arms: Traditional (Standard) Protocol
Drug: Meloxicam — meloxicam tablet
  Other Names: mobic
  Arms: Multimodal Anesthesia and Analgesia

SUMMARY:
Opioid medications are associated with many side effects and the risk of abuse or overdose. Orthopaedic surgeons are currently investigating ways to control pain after surgery while limiting the amount of opioid medications prescribed. One way to reduce the amount of opioid medications prescribed, and potentially avoid opioid-associated adverse events, is to use multiple non-opioid medications and anesthetic drugs before surgery, during surgery, and after surgery. This study aims to evaluate a protocol with non-opioid pain medications to reduce the need for opioid medication after shoulder surgery.

DETAILED DESCRIPTION:
The United States constitutes <5% of the world's population but over 80% of the opioid supply and 99% of the hydrocodone supply. In 2014, there were 18,893 deaths from prescription drug overdose, and orthopaedic surgeons are the third highest prescribing physicians for opioids. Surgeons often prescribe opioids to minimize postoperative pain and to reduce the likelihood of readmission for pain. Available data suggests that orthopaedic surgeons are the most likely physicians to prescribe opioids to Medicare patients. Among Medicare patients, opioid prescriptions are over 7 times more likely to come from an orthopaedic surgeon than another type of physician. Yet, despite the significant amount of opioids prescribed by orthopaedic surgeons, orthopaedic surgeons often have one of the highest readmission rates for post-operative pain. Many studies have investigated the utilization of opioids after surgery to assess surgeon's tendencies to overprescribe, demographics of those likely to overuse, and adverse events of opioid abusers.

A recent paper by Kim et al. prospectively investigated opioid utilization after upper extremity surgery. This study (n=1,416) showed an opioid utilization rate of just 34%, taking an average 8.1 pills out of 24 prescribed. Patients aged 30-39, those having joint procedures, upper extremity/shoulder surgery, or self-pay/Medicaid insurance were all far more likely to overuse opioids. The study concluded that their surgeons prescribed 3 times the required opioid following surgery and gave recommendations for opioid distribution based on location, procedure type, and patient risk factors. This study's identification of over prescription is congruent with a study completed by Bates et al that showed 67% of patients had a surplus of medications, with 92% not receiving proper medication disposal instructions.

Other recent literature has attempted to risk stratify patients who are more likely to abuse prescription opioids. Morris et al. identified various risk factors including: family history of substance abuse, nicotine dependency, age <45, psychiatric disorders, and lower level of education.These risk factors are associated with aberrant behaviors (non-compliance, early refill request, "lost or stolen" medication), which should raise concerns for any provider prescribing opioids.

Studies have shown that patients who are on chronic opioid therapy before surgery have worse outcomes. A recent study compared chronic opioids users (n= 35,068) versus those who were opioid-naïve at the time of total knee arthroplasty (TKA) and found the opioid group had more opioid scripts filled per patient at discharge as well as at 3, 6, and 9 months (0.63 scripts/patient vs. 1.2 scripts/patient, p<0.05). These patients also had a higher Charlson Comorbidity Index (p<0.05) and higher rates of respiratory failure, acute kidney failure, pneumonia, all post-operative infections, and infections requiring return to the OR. The study concluded patients should have their opioid consumption controlled during the pre-operative and peri-operative period.

In addition to the complications of opioid medications experienced by orthopaedic patients, a recent nationwide retrospective analysis presents an unintended yet severe problem associated with opioid prescriptions. The incidence of pediatric hospitalizations for opioid toxicity nearly tripled from 1997 to 2012. The over-prescription of opioids creates a readily available source for accidental ingestion by younger children and for intentional opioid overdose by older pediatric/adolescent patients. In fact, a family member's leftover pills have been described as the number one source for pediatric opioid overdose. Moreover, the Center for Disease Control reported that in 2015 the U.S. saw its highest incidence of opioid-related death. Given the frequency and severity of opioid diversion and misuse, orthopaedic surgeons should consider the best methods for controlling patients postoperative pain and also avoid facilitating opiate misuse, whether by orthopaedic patients or other community members. With this goal in mind, this study will investigate regimens for effective postoperative pain control that also minimize the total amount of opioids prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of Age, undergoing primary anatomic or reverse total shoulder arthroplasty

Exclusion Criteria:

* Opioid consumption within 4 weeks prior to surgery, allergy to oxycodone or study drugs, refusal to take oxycodone or study drugs, history of opioid dependence or illegal/"off-label" opioid use, revision arthroplasty procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Oxycodone tablets | From time of discharge until the date the subject is no longer using oxycodone or up 90 days after surgery, whichever came first
  Number of tablets taken by patient after hospital discharge

SECONDARY OUTCOMES:
Patient Reported Outcome Measures | administered preoperatively, 6 weeks, 3 months
  Standard shoulder surveys assessing activity and pain
Shoulder range of motion and strength testing | tested as appropriate at 3 weeks, 6 weeks, and 3 months
  postoperative shoulder range of motion and strength testing
Complications | Up to 90 days
  Deep vein thrombosis, pulmonary embolism, return to surgery, hospital readmission, superficial or deep infection, periprosthetic fracture, cerebrovascular accident or transient ischemic attack, dislocation, and opioid withdrawal
Pain Score | From time of randomization until the date of hospital discharge, assessed up to 90 days after surgery.
  Inpatient Pain Score- Visual Analog Scale (VAS) for pain. This is a standard pain evaluation scale rating pain 0 (no pain) to 10 (worst imaginable pain). Lower scores indicate a better outcome.
Postoperative Inpatient Opioid Utilization | From time of randomization until the date of hospital discharge, assessed up to 90 days after surgery.
  Amount of opioid medications taken by patient in hospital
Long-term Pain Scores | Assessed on a weekly basis from the time of discharge up to 90 days after surgery.
  Pain scores of patient after hospital discharge- Visual Analog Scale (VAS) for pain. This is a standard pain evaluation scale rating pain 0 (no pain) to 10 (worst imaginable pain). Lower scores indicate a better outcome.

OTHER OUTCOMES:
Illinois Prescription Monitoring Program (IPMP) | Up to 90 days
  Patient compliance with IPMP

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P Nicholson, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630
- [Background] Morris BJ, Mir HR. The opioid epidemic: impact on orthopaedic surgery. J Am Acad Orthop Surg. 2015 May;23(5):267-71. doi: 10.5435/JAAOS-D-14-00163. PMID 25911660
- [Background] Bates C, Laciak R, Southwick A, Bishoff J. Overprescription of postoperative narcotics: a look at postoperative pain medication delivery, consumption and disposal in urological practice. J Urol. 2011 Feb;185(2):551-5. doi: 10.1016/j.juro.2010.09.088. Epub 2010 Dec 18. PMID 21168869
- [Background] Gaither JR, Leventhal JM, Ryan SA, Camenga DR. National Trends in Hospitalizations for Opioid Poisonings Among Children and Adolescents, 1997 to 2012. JAMA Pediatr. 2016 Dec 1;170(12):1195-1201. doi: 10.1001/jamapediatrics.2016.2154. PMID 27802492
- [Background] Moreno MA. Page for patients. The misuse of prescription pain medicine among children and teens. JAMA Pediatr. 2015 May;169(5):512. doi: 10.1001/jamapediatrics.2014.2128. No abstract available. PMID 25938654
- [Background] Della Valle CJ, Dittle E, Moric M, Sporer SM, Buvanendran A. A prospective randomized trial of mini-incision posterior and two-incision total hip arthroplasty. Clin Orthop Relat Res. 2010 Dec;468(12):3348-54. doi: 10.1007/s11999-010-1491-5. Epub 2010 Jul 29. PMID 20668969
- [Background] Namdari S, Nicholson T, Abboud J, Lazarus M, Steinberg D, Williams G. Randomized Controlled Trial of Interscalene Block Compared with Injectable Liposomal Bupivacaine in Shoulder Arthroplasty. J Bone Joint Surg Am. 2017 Apr 5;99(7):550-556. doi: 10.2106/JBJS.16.00296. PMID 28375887
- See also: Opioid Addiction Facts and Figures 2016 from the American Society of Addiction Medicine — https://www.asam.org/docs/default-source/advocacy/opioid-addiction-disease-facts-figures.pdf
- See also: Opioid Use, Misuse, and Abuse in Orthopaedic Practice from the American Academy of Orthopaedic Surgeons — https://www.aaos.org/uploadedFiles/PreProduction/About/Opinion_Statements/advistmt/1045%20Opioid%20Use,%20Misuse,%20and%20Abuse%20in%20Practice.pdf
- See also: White House Report-Continued Rise in Opioid Overdose Deaths in 2015 Shows Urgent Need for Treatment — https://obamawhitehouse.archives.gov/the-press-office/2016/12/08/continued-rise-opioid-overdose-deaths-2015-shows-urgent-need-treatment

DOCUMENTS (1):
  • Informed Consent Form (2018-09-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT03586934/ICF_000.pdf